CLINICAL TRIAL: NCT06280365
Title: Effects of Mulligan Mobilization With Movement (MWM) Technique in Patients With Knee Osteoarthritis
Brief Title: MWM Technique in Patients With Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Mobilization
Keywords: Knee Osteoarthritis; Mobilization; Proprioception; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWM group (Experimental): Participants in group 2 will receive MWM technique treatment 3 times a week for 4 weeks. The patient should lie face down with a pillow over the knee and the physiotherapist should stand on the contralateral side for the application. The physiotherapist passes the belt around the waist to the patient's tibia edge. The knee is stabilized with one hand while the leg is supported with the other hand. The knee is moved medially without applying too much force through the belt and the patient is asked to stretch. If there is no pain, the movement is indicated. If pain occurs during the movement, the same procedure is performed for the lateral side by changing the position. It is important that the arch remains horizontal and does not cause rotation of the hip. The movement will be repeated 3 times at the point where there is no pain.
  Interventions: Other: Mulligan Mobilization with Movement Technique
- Control Group (No Intervention): Participants in group 1 will receive conservative treatment 3 times a week for 4 weeks. Conservative treatment includes hot packs and traditional transcutaneous electrical nerve stimulation (TENS), an electrotherapy.
  All participants in the study will receive 20 minutes of hot pack application to the knee area each session by a physiotherapist. All participants in the study will receive TENS for 20 minutes each session from the physiotherapist, who will place personalized electrodes around the knee joint and adjust the current to the level the person can tolerate.

INTERVENTIONS:
Other: Mulligan Mobilization with Movement Technique — Mobilization Technique
  Arms: MWM group

SUMMARY:
The aim of this study is to investigate the effect of the MWM technique on pain, normal joint movement, proprioception and quality of life in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of the MWM technique on pain, normal joint movement, muscle strength, proprioception, mobility, balance, functionality and quality of life in patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with knee osteoarthritis,
* being diagnosed with knee OA at the earliest 6 months ago

Exclusion Criteria:

* Participants who were pregnant,
* had knee surgery, had an infection,
* had a pacemaker, had an infraction,
* had cancer, or were receiving corticosteroid treatment were excluded from the study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 week change in pain intensity
  VAS, which digitizes parameter values that cannot be measured numerically, was used to evaluate the pain intensity of the participants. The two extreme values of the parameter to be measured are written on the scale as 0 and 10. The person is asked to mark the value that best suits him/her on the scale. For pain, no pain and very severe pain; It is specified as 0 and 10. The person chooses a value according to his/her pain
Short form-36 (SF-36) | 4-week change in quality of life
  SF-36, developed in 1992, consists of 36 items providing measurement to the following 8 dimensions: physical functioning (10 items), social functioning (2 items), role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items), and general health perception (5 items). An increase in the score indicates a higher rate of improvement in health status.
Western Ontario and Mcmaster Universities Osteoarthritis Index (WOMAC) | 4-week
  This survey is conducted to evaluate how much the routine activities in the participants' lives are affected by the knee problem. The survey included the following parameters: pain, physical function, and stiffness. A Likert system ranging from 1 to 5 is used. As the value increases, the intensity of the parameters increases
Evaluation of proprioception | 4-week change in proprioception
  To assess the participants' sense of proprioception, the method of actively reproducing the passive position without supporting the limb was used. In this assessment, where the angle is measured with a goniometer, the person closes their eyes. The limb is passively moved to the target angle and the person is asked to concentrate on the position. After 10 seconds, the starting point of the movement is returned. The person tries to find the target angle by actively moving the same limb. If the angle achieved at the end of the movement is different from the target angle, the difference is recorded as the deviation angle (used to 15° and 45° knee flexion).
The range of motion | 4-week
  A goniometer (Baseline plastic goniometer), which provides numerical and objective results, was used to measure the range of motion of the participants. Knee flexion for normal range of motion in the knee region and knee extension angles were evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Atıcı, Tuzla, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No